CLINICAL TRIAL: NCT01432652
Title: Efficacité du Traitement antiagrégant Par Acide acétylsalicylique en Chirurgie Vasculaire mesurée Par agrégométrie Par impédance
Brief Title: The Efficacy of Aspirin in the Postoperative Period in Vascular Surgery
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Other Study IDs: 176/11
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2011-09

CONDITIONS: Aspirin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vascular surgery: Patients undergoing vascular surgery

SUMMARY:
The purpose of this study is to determine the incidence of aspirin resistance in the population of vascular surgery patients; and to evaluate the changes in the efficacy of aspirin in the first five postoperative days.

DETAILED DESCRIPTION:
About 15% of the general population shows resistance to the antiplatelet effects of aspirin, due to genetic polymorphisms and other factors. This resistance is a cause of increased myocardial infarction and death in patients undergoing percutaneous coronary interventions. Aspirin resistance can be detected by whole blood impedance aggregometry using the Multiplate® analyzer. The population of patients undergoing vascular surgery is at particular risk of suffering myocardial infarction in the perioperative period because of the high prevalence of risk factors. Most of these patients are treated by aspirin, as a measure of primary or secondary prevention. In this study we aim to establish baseline aspirin efficacy, as measured by the Multiplate® analyzer, in this high-risk population and evaluate the changes in aspirin efficacy over the first five days of the postoperative period. It is our hypothesis that the state of chronic inflammation, accompanying severe, generalized atherosclerosis results in a higher incidence of aspirin resistance in this population. Also, the surgical trauma and postoperative thrombocytosis may reduce the efficacy of aspirin in the postoperative period, partially explaining the increased incidence of postoperative myocardial infarction in this population.

In whole blood impedance aggregometry, the electrical impedance of the blood sample is measured by placing two electrodes in the recipient. After the addition of a platelet activator, the impedance will increase as platelets accumulate on the electrodes surfaces. Several activators, testing the patency of different platelet receptors can be used.

In this study, blood will be drawn on the day of surgery, and daily until the fifth postoperative day. Arachidonic acid, ADP, TRAP-6 and collagen will be used as activators. The first specifically tests the platelets reactivity to thromboxane A2. Aspirin inhibits this pathway, and the increase in impedance should therefore be limited in patients treated by this drug. The three other tests will be performed to evaluate the evolution of overall platelet reactivity in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing peripheral vascular or abdominal aorta surgery.
* Patient aged 18 years or older.
* Patient treated by aspirin.

Exclusion Criteria:

* Incapacity to understand and consent to study.
* Patient undergoing emergency surgery.
* Patient treated by a cox-inhibitor other than aspirin.
* Patient treated by omega-3-fatty acids.
* Patient treated by ADP or GPIIb/IIIa receptor inhibitor.
* Known coagulopathy, thrombopenia, thrombopathia or congenital or acquired thrombasthenia.
* Terminal renal insufficiency.
* Hepathic insufficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vascular surgery patients
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland